CLINICAL TRIAL: NCT05965934
Title: A Prospective, Randomized Study of Infusate 2.0 Direct Sodium Removal (DSR) Treatment in Subjects With Chronic Heart Failure (CHF) Induced Persistent Congestion, Resistant to Loop Diuretic Treatment.
Brief Title: Management of Volume Overload HF Patients by Individual DSR Treatment adJustment-a clinicAl inVestigation of InfusatE2.0
Acronym: MOJAVE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-CHF-012
Record Dates: First submitted 2023-07-13; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Volume Overload
Keywords: Direct Sodium Removal
MeSH Terms: conditions — Heart Failure; Edema | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Direct Sodium Removal (DSR) Infusate 2.0 (Experimental): Participants will receive a peritoneal dialysis catheter implant. DSR is to be started 14 days after catheter implantation (= D1) for a period of 4 weeks (D28) on top of optimized usual care for HF, while loop diuretic treatment is suspended. Participants then enter enter a 3 month safety follow-up period (D29-D120) until the end of study (D120).
  Interventions: Drug: Direct Sodium Removal Infusate 2.0
- Optimized Usual Care for HF (No Intervention): IV loop diuretic treatment is to be started (or continued) after a 14 days observation period (= D1) and can be continued for up to 4 weeks (D28). Participants then enter enter a 3 month safety follow-up period (D29-D120) until the end of study (D120).

INTERVENTIONS:
Drug: Direct Sodium Removal Infusate 2.0 — Direct Sodium Removal via peritoneal ultrafiltration using Infusate 2.0 (30% icodextrin, 10% dextrose). Patients (if not yet on SGLT-2 inhibitors) will receive SGLT-2 inhibitors.
  Other Names: SGLT-2 inhibitor (dapagliflozin)
  Arms: Direct Sodium Removal (DSR) Infusate 2.0

SUMMARY:
This study is a multi-center, prospective, randomized (2:1), open-label study to evaluate the safety and efficacy of DSR therapy using the Infusate 2.0 peritoneal solution (composed of 30% icodextrin and 10% dextrose) in diuretic resistant patients with HF and persistent volume overload.

DETAILED DESCRIPTION:
The study will start with a non-randomized cohort in which 3 eligible subjects will be treated with Infusate 2.0 on top of their usual care while all loop diuretic treatment is stopped. A Peritoneal Dialysis (PD) catheter will be implanted to administer the infusate 14 days post-PD catheter implantation. The infusate will be drained via the same route after up to 24 hr dwell time. This DSR process will be repeated up to daily over a treatment period of 4 weeks (D1-D28). The quantity of infusate and the duration of dwell time will be adjusted based on treatment effect and tolerability.

After the treatment period, the PD catheter is removed and a 3 month safety follow-up period starts to the end of study (D29-D120).

After Data and Safety Monitoring Board (DSMB) review of 30 days follow-up data (D58) of the non-randomized cohort and DSMB approval to proceed, the 2:1 randomized enrollment of up to 30 additional subjects will be opened.

* DSR Group (N = 20) Treatment: DSR Infusate 2.0 DSR is to be started 14 days post-PD catheter implantation (= D1) for a period of 4 weeks (D28) on top of optimized usual care for HF, while loop diuretic treatment is suspended.
* Control Group (N = 10) Treatment: Optimized usual care for HF IV loop diuretic treatment is to be started (or continued) after a 14 days observation period (= D1) and can be continued for up to 4 weeks (D28).

All subjects should then enter the 3 month safety follow-up period (D29-D120) until the end of study (D120).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at screening
* Weight at screening ≥50 kg (110 lbs)
* Creatinine-based estimated glomerular filtration rate (eGFR) (CKD-EPI] 2021 formula) ≥30 mL/min/1.73m² at screening
* 6-hour cumulative urine sodium excretion <100 mmol to 40 mg IV furosemide on diuretic challenge
* Diagnosis of symptomatic heart failure with NYHA class III or IV AND daily diuretic dose ≥80 mg furosemide (or ≥20 mg torsemide or ≥1 mg bumetanide) for ≥14 days prior to screening AND NT-proBNP >2000 pg/mL (or BNP >400 pg/mL) OR oral daily diuretic dose ≥160 mg furosemide (or ≥40 mg torsemide or ≥2 mg bumetanide) over the previous 14 days AND ≥2 HF volume overload events within the last 6 months prior to screening or 2 HF volume overload-related hospitalizations within the last 12 months prior to screening
* Persistent mild to moderate volume overload with ≥2,3 kg (5 lbs) of excess hypervolemia AND more than trace peripheral edema AND/OR jugular venous distention AND/OR elevated filling pressure on chronic remote pressure monitoring device
* Systolic blood pressure ≥90 mmHg and <180 mmHg
* Receiving maximally tolerated stable doses of guideline-directed medical therapy (GDMT)
* For participants of childbearing potential: negative pregnancy test and agreement to use highly effective contraception for ≥1 month prior to screening and until ≥3 months after last exposure to investigational medicinal product
* For participants with intimate partners of childbearing potential: agreement to use highly effective contraception for ≥1 month prior to screening and until ≥3 months after last exposure to investigational medicinal product

Exclusion Criteria:

* Reversible cause of persistent decompensation or diuretic resistance
* Contraindications for peritoneal dialysis (PD) or PD catheter placement
* Known contraindication to icodextrin use
* Known contraindication or intolerance or allergy to SGLT2 inhibitors
* Current diagnosis of severe bladder dysfunction
* Imminent need for hospitalization
* Current or prior (past 6 months) use of renal replacement therapy
* Anemia with hemoglobin <8 g/dL
* Serum sodium <130 mEq/L
* Severe albuminuria (urinary albumin/creatinine ratio >1 at screening)
* Severe cardiac cachexia
* Clinically significant cirrhosis or history of clinically significant ascites (i.e., prior large volume paracentesis) or large volume ascites on imaging or exam
* Type 1 diabetes, uncontrolled Type 2 diabetes, "brittle" diabetes or frequent hypoglycemia or severe hyperglycemic episodes requiring emergent intervention in the last 6 months
* Known or suspected low output HF
* Prior or planned heart transplant or mechanical cardiac support implantation (LVAD)
* History of severe hyperkalemia > 5.5 mEq/L (past 6 months) or screening plasma potassium >4.5 mEq/L
* Significant non-cardiac disease or comorbidities expected to reduce life expectancy to <1 year or to interfere with safety or conduct of the study
* Severe restrictive or obstructive HF or hemodynamically significant, severe uncorrected stenotic valvular disease
* Receiving anticoagulation or antiplatelet treatment, which cannot be withheld (bridging therapy allowed)
* Recent myocardial infarction, cerebrovascular accident, transient ischemic attack, coronary revascularization, arrhythmia ablation, cardiac resynchronization therapy, or surgical or transcatheter valve intervention (within 90 days prior to screening)
* Received treatment with other investigational products or devices within 30 days of screening or 5 halflives of the previous investigational product
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate through end of treatment period | from Day 1 to day 28 (treatment period)
  Safety
Serious adverse event rate through end of treatment period | from Day 1 to day 28 (treatment period)
  Safety

SECONDARY OUTCOMES:
Change in Urine sodium output from baseline to end of treatment period | from Day 1 to day 28 (treatment period)
  Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Turner, MD, Principal Investigator — Yale Universtiry; Marath Fudim, MD MHS, Principal Investigator — Duke University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] McIntyre CW. Update on Hemodialysis-Induced Multiorgan Ischemia: Brains and Beyond. J Am Soc Nephrol. 2024 May 1;35(5):653-664. doi: 10.1681/ASN.0000000000000299. Epub 2024 Jan 26. PMID 38273436